CLINICAL TRIAL: NCT07311408
Title: SHR-1701 Combined With Rivoceranib, With or Without SHR-2554, in Patients With Advanced Gastric Cancer Who Have Failed First-Line Immunotherapy
Brief Title: SHR-1701 + Rivoceranib (± SHR-2554) in Advanced GC After First-Line Immunotherapy Failure
Acronym: SHR-2554
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jingdong Zhang (Other)
Responsible Party: Sponsor-Investigator, Jingdong Zhang, Chief Physician, Professor, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-029; will be entered later (Other Grant/Funding Number: will be entered later)
Record Dates: First submitted 2025-11-30; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer (GC); Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Rivoceranib; Failed First-Line Immunotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — SHR-1701; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1701+Rivoceranib + SHR-2554 (Experimental): Drug: SHR-1701 Administered by intravenous (IV) infusion on Day 1 of each 21-day cycle. The infusion time should be controlled between 30 and 60 minutes, and must not exceed 2 hours.
  Drug: Rivoceranib Administered orally (PO) once daily (QD), continuously. Administration Instructions: To be taken orally with warm water, approximately 30 minutes after a meal. The daily dosing time should be consistent.
  Drug: SHR-2554 Administered orally (PO) twice daily (BID). Administration Instructions: Can be taken before or after meals, but administration approximately 30 minutes after morning and evening meals is recommended. The daily dosing times should be consistent.
  Interventions: Drug: SHR-1701 + Rivoceranib
- SHR-1701 + Rivoceranib. (Active Comparator): Drug: SHR-1701 Administered by intravenous (IV) infusion on Day 1 of each 21-day cycle. The infusion time should be controlled between 30 and 60 minutes, and must not exceed 2 hours.
  Drug: Rivoceranib Administered orally (PO) once daily (QD), continuously. Administration Instructions: To be taken orally with warm water, approximately 30 minutes after a meal. The daily dosing time should be consistent.
  Interventions: Drug: SHR-1701+Rivoceranib + SHR-2554

INTERVENTIONS:
Drug: SHR-1701+Rivoceranib + SHR-2554 — Drug: SHR-1701 Administered by intravenous (IV) infusion on Day 1 of each 21-day cycle. The infusion time should be controlled between 30 and 60 minutes, and must not exceed 2 hours.
  Drug: Rivoceranib Administered orally (PO) once daily (QD), continuously. Administration Instructions: To be taken orally with warm water, approximately 30 minutes after a meal. The daily dosing time should be consistent.
  Drug: SHR-2554 Administered orally (PO) twice daily (BID). Administration Instructions: Can be taken before or after meals, but administration approximately 30 minutes after morning and evening meals is recommended. The daily dosing times should be consistent.
  Arms: SHR-1701 + Rivoceranib.
Drug: SHR-1701 + Rivoceranib — Drug: SHR-1701 Administered by intravenous (IV) infusion on Day 1 of each 21-day cycle. The infusion time should be controlled between 30 and 60 minutes, and must not exceed 2 hours.
  Drug: Rivoceranib Administered orally (PO) once daily (QD), continuously. Administration Instructions: To be taken orally with warm water, approximately 30 minutes after a meal. The daily dosing time should be consistent.
  Arms: SHR-1701+Rivoceranib + SHR-2554

SUMMARY:
To investigate the efficacy of SHR-1701 combined with Rivoceranib, with or without SHR-2554, in patients with gastric or gastroesophageal junction adenocarcinoma who have progressed on or were intolerant to first-line immunotherapy-containing treatment

DETAILED DESCRIPTION:
This is a prospective, open-label, dual-cohort, Phase II clinical study designed to observe and evaluate the efficacy and safety of SHR-1701 combined with Rivoceranib, with or without SHR-2554, in patients with advanced gastric cancer who have failed first-line immunotherapy. The study targets patients with gastric or gastroesophageal junction adenocarcinoma who have progressed on or are intolerant to first-line immunotherapy-containing regimens. Eligible subjects who provide informed consent and pass screening will be randomized in a 1:1 ratio to receive the study treatment.

Cohort 1: SHR-1701+ Rivoceranib+ SHR-2554；Cohort 2: SHR-1701 + Rivoceranib. Primary Endpoint (based on RECIST v1.1): Progression Free Survival (PFS); Secondary Endpoints (based on RECIST v1.1): Objective Response Rate (ORR); Duration of Response (DoR); Overall Survival (OS); Safety; Exploratory Endpoint: Multi-omics analysis of the tumor microenvironment (including, but not limited to, ctDNA and TMB).

Official Title：A Prospective, Dual-Cohort, Phase II Clinical Study of SHR-1701 Combined with Rivoceranib With or Without SHR-2554 in Patients with Advanced Gastric Cancer Who Failed First-Line Immunotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female.
2. Histologically or pathologically confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma.
3. Disease progression on or intolerance to a prior treatment regimen that contained an immune checkpoint inhibitor (ICI).
4. HER2-negative expression.
5. Willingness to provide tumor tissue samples from prior to the first systemic therapy for biomarker analysis (e.g., PD-L1). Freshly obtained biopsies are preferred; if unavailable, archived formalin-fixed paraffin-embedded (FFPE) tissue blocks or 5-8 slides of 3-5μm thickness are acceptable.
6. At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Life expectancy ≥ 12 weeks.
9. Adequate organ and bone marrow function, defined as:

   1. Hemoglobin ≥ 90 g/L (no blood transfusion within 14 days);
   2. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   3. Platelet count ≥ 90 × 10^9/L;
   4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN);
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; for patients with liver metastases, ALT and AST ≤ 5 × ULN;
   6. Serum creatinine ≤ 1.5 × ULN;
   7. Left ventricular ejection fraction (LVEF) ≥ 50%; QTc interval < 450 ms for males and < 470 ms for females.
10. For patients not on therapeutic anticoagulation: International Normalized Ratio (INR) ≤ 1.5 and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN. Patients receiving full-dose or parenteral anticoagulants are eligible provided the dose has been stable for at least 2 weeks prior to study entry and relevant coagulation parameters are within the therapeutic range.
11. For women of childbearing potential: a negative serum or urine pregnancy test within 14 days prior to enrollment, and agreement to use highly effective contraception during the study and for 3 months after the last dose of the study drug. For male patients: surgical sterilization or agreement to use highly effective contraception during the study and for 3 months after the last dose.
12. Recovery from toxicities of prior therapies to ≤ Grade 1 (per NCI CTCAE). For prior surgeries, the wound must have healed completely.
13. Voluntary participation, provision of signed informed consent, expected good compliance, and ability to comply with the study protocol requirements.

Exclusion Criteria:

1. Gastrointestinal perforation and/or fistula within 6 months prior to treatment, or active gastrointestinal bleeding within 3 months.
2. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
3. Known history of allergy to any component of the investigational drugs or their excipients.
4. Prior treatments as follows:

   1. Treatment with any other investigational agent within 4 weeks prior to the first dose of the study drug, or within 5 half-lives of the previous investigational agent (whichever is longer).
   2. Concurrent enrollment in another interventional clinical study. (Observation studies or follow-up phases of interventional studies are permitted).
   3. Any antitumor therapy (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biotherapy, or tumor embolization) within 2 weeks prior to the first dose of the study drug.
   4. Requirement for systemic corticosteroids (>10 mg prednisone equivalent daily) within 2 weeks prior to the first dose. The use of corticosteroids for premedication with certain chemotherapy regimens, inhaled or topical steroids, and adrenal replacement therapy at doses ≤10 mg/day prednisone equivalent is permitted. Other cases require discussion with the Investigator.
   5. Prior administration of an anti-tumor vaccine or live vaccine within 4 weeks prior to the first dose.
   6. Major surgery or significant trauma within 4 weeks prior to the first dose.
5. History of leptomeningeal metastasis, or current evidence of leptomeningeal metastasis or active brain metastases. (Patients with stable, treated brain metastases may be discussed for eligibility).
6. Active autoimmune disease or history of autoimmune disease requiring systemic treatment in the past 2 years. Exceptions include vitiligo, resolved childhood asthma/atopy, hypothyroidism stable on hormone replacement, or Type I diabetes stable on insulin regimen.
7. Immunodeficiency history, including positive HIV test, other acquired/congenital immunodeficiency disorders, history of organ transplant or allogeneic bone marrow transplantation, or active hepatitis.
8. Poorly controlled cardiovascular diseases, including but not limited to: (1) Heart failure of NYHA Class II or higher; (2) Unstable angina; (3) Myocardial infarction within the past year; (4) Clinically significant supraventricular or ventricular arrhythmia without effective medical control.
9. Severe infection within 4 weeks prior to the first dose. Active pulmonary inflammation on baseline imaging, or signs/symptoms of active infection within 2 weeks prior to the first dose.
10. History of interstitial lung disease.
11. Active tuberculosis infection based on history/CT findings, or history of active TB within one year prior to enrollment, or prior active TB over one year ago without appropriate treatment.
12. Diagnosis of another malignancy within 5 years prior to the first dose. Exceptions include malignancies with low risk of metastasis/death.
13. Pregnancy or lactation.
14. Any other condition deemed by the investigator to potentially compromise patient safety or study compliance. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the date of first treatment until the date of first documented disease progression (assessed per RECIST 1.1) or death from any cause, whichever occurs first, assessed up to 24 months.
  To evaluate the efficacy of anti-tumor by Resist1.1 (In months)

SECONDARY OUTCOMES:
Objective response rate (ORR) | From the start of treatment until the first occurrence of documented complete response (CR) or partial response (PR) per RECIST 1.1, assessed up to 24 month
  To evaluate the efficacy of anti-tumor by Resist1.1
Disease control rate (DCR) | From the start of treatment until the first documented complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1, assessed up to 24 months.
  To evaluate the efficacy of anti-tumor by Resist 1.1 (In percent)
Overall survival (OS) | From the date of first treatment until the date of death from any cause, assessed up to 36 months
  To evaluate the efficacy of anti-tumor by Resist 1.1 (In months)
Safety | From the first dose of study treatment until 30 days after the last dose, assessed up to approximately 26 months.
  Incidence and severity of treatment-emergent adverse events (TEAEs).

OTHER OUTCOMES:
Multi-omics analysis of the tumor microenvironment | From enrollment to the end of the study
  ctDNA, TMB, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Provincial Cancer Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided